CLINICAL TRIAL: NCT03614065
Title: Endostar Combine With Radiotherapy in Brain Metastasis of NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaorong Dong, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: endobrain
Record Dates: First submitted 2016-08-08; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — endostar protein; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm a (Placebo Comparator): This group is a placebo control group, and we will use radiation therapy plus Placebos as the control group for the study
  Interventions: Drug: Placebos; Radiation: radiotherapy
- arm b (Experimental): This group belongs to the experimental group. We will use radiotherapy combined with endostar for treatment, so as to judge the efficacy of the medicine
  Interventions: Drug: endostar; Radiation: radiotherapy

INTERVENTIONS:
Drug: endostar — endostatin
  Other Names: An antiangiogenic drug
  Arms: arm b
Drug: Placebos — saline solution
  Other Names: negative control
  Arms: arm a
Radiation: radiotherapy — radiotherapy

SUMMARY:
Observe the effect os radiotherapy plus or not plus endostar in the treatment of brain metastasis in NSCLC

DETAILED DESCRIPTION:
The investigators will observe the time controlled by the brain lesion after the test and the total survival time of the patients. Meanwhile, during each follow-up, the investigators will extract cerebrospinal fluid for genomic analysis of cerebrospinal fluid

ELIGIBILITY:
Inclusion Criteria:

* NSCLC Brain metastasis

Exclusion Criteria:

* KPS<60

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From date of randomization until the date of first documented progression of brain lesions, and the maximum evaluation time is 36 months
  the time from the start of treatment to the progression of the brain metastases, in months

SECONDARY OUTCOMES:
Overall survival （OS） | From date of randomization until the date of death, assessed up to 36 months
  the total survival time of the patient from the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: dong xiaorong, Dr, Study Director — china goverment
Locations (1):
- Union Hospital, Wuhan, Hubei, China